CLINICAL TRIAL: NCT01660633
Title: A Phase IIb, Multicenter, Open-Label, Safety and Efficacy Study of High Dose Melphalan HCL for Injection (Propylene Glycol-Free)for Myeloablative Conditioning in Multiple Myeloma Patients Undergoing Autologous Transplantation
Brief Title: Safety & Efficacy Study High Dose Evomela Injection for MA Conditioning in MM Patients With Autologous Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Acrotech Biopharma Inc. (Industry)
Collaborators: Clinipace Worldwide (Industry); Beckloff Associates, Inc. (Industry); Kansas City Bioanalytical Laboratories (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDX-353-002
Record Dates: First submitted 2012-08-02; First posted 2012-08-09 (Estimated); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; High-Dose Melphalan; Propylene Glycol-Free; Autologous Stem Cell Transplantation; Captisol
MeSH Terms: conditions — Multiple Myeloma | interventions — Melphalan; Injections; Transplantation, Autologous; Hematopoietic Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- High-Dose Melphalan HCL for Injection (Propylene Glycol-Free) (Other): Subjects will receive only High-Dose Melphalan HCL for Injection (Propylene Glycol-free) at 200mg/m2 (100mg/m2/day for two days).
  Interventions: Drug: High-Dose Melphalan HCL for Injection (Propylene Glycol-Free); Other: Autologous Transplantation

INTERVENTIONS:
Drug: High-Dose Melphalan HCL for Injection (Propylene Glycol-Free) — 200 mg melphalan/m2 will be divided into two separate, consecutive doses of 100 mg/m2 administered on day -3 and day -2 prior to ASCT. The High-Dose Melphaln HCL for Injection (Propylene Glycol-Free) will be reconstituted to 5 mg/mL (also containing 270 mg/mL of Captisol®). The Melphalan HCL for Injection (Propylene Glycol Free) will be further diluted with normal saline to a concentration of no greater than 0.45 mg/mL and infused over 30 minutes ( + or - 3 minutes)via a central venous catheter.
  Other Names: Evomela; Alkeran
Other: Autologous Transplantation — Patients who are myeloablative conditioning in multiple myeloma undergoing autologous transplantation( patients own blood-forming stem cells are collected to replace diseased bone marrow or bone marrow damaged by cancer treatment)
  Other Names: Hematopoietic stem cell transplantation

SUMMARY:
The purpose of this trial is to confirm the safety and efficacy of high-dose Melphalan HCL for Injection (Propylene Glycol-Free) as a myeloablative conditioning regimen in multiple myeloma patients (MM) undergoing autologous transplantation.

DETAILED DESCRIPTION:
The sponsor of the current study is now Acrotech Biopharma, divested from Spectrum Pharmaceuticals Inc. (Spectrum), which licensed the Melphalan HC1 for Injection (Propylene Glycol-Free) product from Ligand Pharmaceuticals , formerly CyDex Pharmaceuticals, Inc. (CyDex). This new injectable form of melphalan HCL incorporates Captisol®, β cyclodextrin sulfobutyl ether sodium salts (also known as [SBE]7m-β-CD), into the product. Captisol is present to facilitate the use of an all aqueous diluent (normal saline) for reconstitution and administration of the freeze-dried product in place of the propylene glycol-ethanol diluent necessary for the currently used melphalan intravenous product. Captisol provides for solubilization and improved stability of the all aqueous reconstituted and diluted infusion solution.

This is the second of two studies supporting product registration. This study will be a multicenter study of high-dose Melphalan HCL for Injection (Propylene Glycol-Free) conducted in 60 patients who have symptomatic MM and qualify for autologous stem cell transplantation (ASCT).

During the Study Period, patients will receive 100mg/m2 of either Melphalan HCL for Injection (Propylene Glycol-Free) on Day -3 and on Day -2 for a total dose of 200mg/m2. Blood samples (5 timepoints post infusion) for population pharmacokinetic (PK) evaluation will be withdrawn through an indwelling i.v. cannula on the first day of administration of melphalan (Day -3) for all patients and then additional blood samples (2 timepoints post infusion) drawn in a subset of patients on the second day of melphalan administration (Day -2).

Following one day of rest after the high dose myeloablative conditioning (Day -1), patients will receive an autologous graft (Day 0).

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic MM based on IMWG guidelines requiring treatment who are eligible for ASCT.
* Patients who are 70 years of age or younger at time of transplant. Patients older than 70 years of age may be enrolled on a case-by-case basis if the patient meets local institutional criteria to receive a total melphalan dose of 200 mg/m2 as a conditioning regimen and if approved by the medical monitor.
* Patients with an adequate autologous graft, defined as an unmanipulated, cryopreserved, peripheral blood stem cell graft containing at least 2 × 106 CD34+ cells/kg based on patient body weight.

Patients with adequate organ function as measured by:

* Cardiac function: Left ventricular ejection fraction at rest >40% (documented within 8 weeks prior to Day -3).
* Hepatic function: Bilirubin <2 × the upper limit of normal and alanine aminotransferase (ALT)/aspartate aminotransferase (AST) <3 × upper limit of normal.
* Renal function: Creatinine clearance >40 mL/minute (measured or calculated/estimated).
* Pulmonary function: Carbon monoxide diffusing capacity (DLCO)corrected for hemoglobin (Hgb), forced expiratory volume in 1 second (FEV1), forced expiratory vital capacity (FVC), and oxygen saturation >92% on room air (documented within 4 weeks prior to Day -3).
* Patients with Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.

Exclusion Criteria:

* Patients with smoldering MM not requiring therapy.
* Patients with plasma cell leukemia.
* Patients with systemic amyloid light chain amyloidosis.
* Patients with uncontrolled hypertension.
* Patients with an active bacterial, viral, or fungal infection.
* Patients with a life expectancy of < 6 months.
* Patients with prior malignancies except resected basal cell carcinoma or treated cervical carcinoma in situ. Cancer treated with curative intent >5 years previously will be allowed. Cancer treated with curative intent <5 years previously will not be allowed unless approved by the medical monitor.
* Female patients who are pregnant or breastfeeding.
* Female patients of childbearing potential who are unwilling to use adequate contraceptive techniques during and for 3 months following study treatment with Melphalan HCl for Injection (Propylene Glycol-Free).
* Patients seropositive for Human Immunodeficiency Virus(HIV).
* Patients who are unwilling to provide informed consent.
* Patients receiving other concurrent anticancer therapy (including chemotherapy, radiation, hormonal treatment, or immunotherapy, but excluding corticosteroids) within 30 days prior to the ASCT or planning to receive any of these treatments prior to Day +30.
* Patients concurrently participating in any other clinical study involving ASCT.
* Patients who are hypersensitive or intolerant to any component of the study drug formulation.

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2012-12; Primary Completion 2014-02 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Up to Day +100
  AE coding will be performed using the MedDRA Version 11.0 or greater. The severity of the toxicities will be graded according to the NCI CTCAE Version 4.0 whenever possible. AEs occurring when treatment starts on Day -3 through Day + 100 will be recorded in the AE section of the eCRF and causality will be assigned by the Principal Investigator.
Mucositis Severity according to World Health Organization Scoring System | Until Day +30
  The baseline measurement will be the last assessment prior to receiving the first dose of study treatment. The on-treatment period will be defined as the day after the first dose of study treatment to 30 days after the last dose of study treatment. The incidence of severe mucositis (WHO Grade 3 or 4) will be summarized by frequencies and percentages. In addition, the incidence of oral mucositis will be summarized by WHO grade. Time from start of the first dose of study medication to peak oral mucositis score will also be calculated.
Mouth Pain Scores according to a Visual Analog Scale | Until Day +30
  Baseline VAS for mouth pain and dysphagia will be the VAS score collected prior to receiving the first dose of study medication. Analyses of changes and/or percent changes from baseline in the VAS scores will be analyzed for each time point collected during the 30 day on-treatment period. The minimum and maximum VAS scores during the 30 day on-treatment period will also be calculated for mouth pain and dysphagia, and the time to the minimum and maximum VAS scores will be summarized descriptively.
Treatment Related Mortality | Up to Day +100
  TRM, which is defined as death not due to disease progression before Day +90/+100, will be calculated. This outcome measure will be summarized by the cumulative incidence estimated with 95% confidence intervals.

SECONDARY OUTCOMES:
MM response according to International Myeloma Working Group (IMWG) criteria. | At the Day +100 visit
  Definition of active MM, clonal bone marrow plasma cells >10% or biopsy-proven bony or extramedullary plasmacytoma and any one or more of the following CRAB features and myeloma-defining events: Evidence of end organ damage that can be attributed to the underlying plasma cell proliferative disorder and one or more biomarkers of malignancy (MDEs) defined in the criteria.
Myeloablation | Up to Day +30
  Absolute neutrophil count (ANC) <0.5 × 109/L, absolute lymphocyte count (ALC) <0.1 × 109/L, platelet count <20,000/mm3, or bleeding requiring transfusion.
Neutrophil engraftment | Up to Day +100
  ANC >0.5 × 109/L × first 3 consecutive daily assessments
Platelet engraftment | Up to Day +100
  Untransfused platelet measurement >20,000/mm3 × first 3 consecutive daily assessments
Non-engraftment | Up to Day +100
  Failure to reach an ANC >0.5 × 109/L × 3 consecutive daily assessments by Day +100.

CONTACTS AND LOCATIONS:
Overall Officials: Tim Freeman, Study Director — Clinipace Worldwide
Locations (6):
- United States (6):
  - Rush University Medical Center, Chicago, Illinois
  - University of Kansas Medical Center, Fairway, Kansas
  - University of Massachusetts, Worcester, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Medical College of Wisconsin/Froedtert Hospital, Milwaukee, Wisconsin